CLINICAL TRIAL: NCT06997822
Title: Integrated Critical Illness Aftercare and Recovery Enhancement (I-CARE) Program
Brief Title: Integrated Recovery Program for Critical Illness
Acronym: iCARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 202502049RINA
Record Dates: First submitted 2025-05-14; First posted 2025-05-30 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-05

CONDITIONS: ICU Survivors
Keywords: ICU survivors; Physical function; Cognitive; Weight loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LINE Bot-Based Remote Care Combined with In-Person Post-ICU Clinic (Experimental): LINE Bot-Based Remote Care includes instructional videos for basic mobility skills, recommended exercise practices, cognitive training, and nutritional education. In addition, survivors can report their signs and symptoms to request relevant educational content. At 3 months, participants will attend a post-ICU clinic for comprehensive assessment, necessary interventions, and care transition planning.
  Interventions: Behavioral: LINE Bot-Based Remote Care Combined with In-Person Post-ICU Clinic
- Non-Interactive LINE Bot + Assessment-Only Clinic (No Intervention): Participants in the control group will be invited to join an official LINE chat, which will not provide any interventions or educational content. They will, however, receive a post-ICU assessment clinic visit at the 3-month follow-up.

INTERVENTIONS:
Behavioral: LINE Bot-Based Remote Care Combined with In-Person Post-ICU Clinic — Participants in this group will receive the I-CARE intervention, which includes two components: (1) a LINE Bot-based remote care system providing scheduled health education, functional assessments, and reminders tailored to ICU survivors, and (2) structured in-person visits to a post-ICU recovery clinic, where multidisciplinary professionals provide follow-up assessments and individualized rehabilitation guidance. The LINE Bot also features an interactive module ("Thanks to Nurses") that allows patients to send messages, images, or audio clips to their ICU care team, with optional reciprocal feedback. The intervention will be delivered for up to 6 months following hospital discharge.
  Arms: LINE Bot-Based Remote Care Combined with In-Person Post-ICU Clinic

SUMMARY:
This study aims to investigate the effects of the Integrated Critical Illness Aftercare and Recovery Enhancement (I-CARE) program on reducing healthcare burden and improving functional outcomes in ICU survivors. The I-CARE program combines remote support via LINE Bot Care with in-person post-ICU recovery clinic visits. The study will assess whether this integrated care model reduces unplanned hospital readmissions and emergency department visits within six months after discharge, and improves physical and cognitive outcomes at 3 and 6 months post-discharge. Additionally, the study will evaluate the impact of a built-in patient-nurse interaction feature on ICU nurses' burnout and intention to leave, measured every six months over a two-year period.

DETAILED DESCRIPTION:
This randomized clinical trial is designed to evaluate the effectiveness of the Integrated Critical Illness Aftercare and Recovery Enhancement (I-CARE) program for survivors of critical illness discharged from the intensive care unit (ICU). The I-CARE program integrates a LINE Bot-based remote monitoring and support system with structured, in-person post-ICU recovery clinic visits. The primary objective is to determine whether this comprehensive care model can reduce the incidence of unplanned hospital readmissions and emergency department visits within six months after hospital discharge.

Secondary outcomes focus on functional recovery and include assessments of physical mobility (e.g., ability to transition from sit to stand), inspiratory muscle strength, body weight changes, presence of dysphagia, and cognitive function at 3 and 6 months post-discharge.

In addition, the LINE Bot Care system incorporates an interactive feature titled "Thanks to Nurses," which enables ICU survivors to share personal reflections, such as short messages, photos, diary entries, stickers, and audio clips, with their ICU care team. This bidirectional communication channel is intended to enhance emotional support and foster a sense of connection between patients and healthcare providers. The study will evaluate the impact of this feature on ICU nurses' professional well-being, specifically measuring levels of burnout and intention to leave the profession at 6, 12, 18, and 24 months after implementation, using a pre-post intervention design.

ELIGIBILITY:
Inclusion Criteria:

* ICU survivors who had experienced endotracheal intubation and mechanical ventilation treatment.

Exclusion Criteria:

* ICU survivors who are unable to walk independently before admission
* ICU survivors who are unable to receive assessment (e.g., dementia or mental retardation)
* ICU survivors who don't have a smartphone.
* ICU survivors were discharged to institutional care facilities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of unplanned hospital readmissions | 1, 2, 3, 4, 5, and 6 months after discharge
Incidence of emergency department visits | 1, 2, 3, 4, 5, and 6 months after discharge

SECONDARY OUTCOMES:
Barthel Index | Immediately after ICU discharge and 0, 3, and 6 months after discharge
  The Barthel Index is a validated instrument used to assess functional independence in activities of daily living (ADLs). It evaluates a person's ability to perform ten basic self-care and mobility tasks, such as feeding, bathing, dressing, grooming, bowel and bladder control, toileting, chair/bed transfers, ambulation, and stair climbing. Scores range from 0 to 100, with higher scores indicating greater independence.
Maximal inspiratory pressure | Immediately after ICU discharge and 0, 3, and 6 months after discharge
  Maximal Inspiratory Pressure (MIP) is a measure of respiratory muscle strength, specifically the strength of the diaphragm and other inspiratory muscles. It is assessed by having the individual inhale as forcefully as possible against an occluded airway, typically measured in centimeters of water pressure (cmH₂O). MIP is a key indicator of ventilatory muscle function and is commonly used in critical care, pulmonary rehabilitation, and neuromuscular disease assessment.
Grip strength | Immediately after ICU discharge and 0, 3, and 6 months after discharge
  Grip strength is a simple and reliable measure of overall muscle strength, particularly of the upper extremities. It is commonly used as a proxy for general physical function and is strongly associated with mobility, nutritional status, and overall health outcomes. Lower grip strength has been linked to increased risk of disability, hospitalization, and mortality.
Modified 30-second sit-to-stand test | Immediately after ICU discharge and 0, 3, and 6 months after discharge
  The Modified 30-Second Sit-to-Stand Test (m30STS) is a functional performance test used to assess lower limb muscle strength and endurance. It measures the number of times an individual can rise from a seated to a standing position in 30 seconds. In the modified version, participants are allowed to use their upper limbs (e.g., pushing off from the chair or armrests) to complete the movement, making it more suitable for frail or physically limited individuals, such as older adults or ICU survivors.
Montreal Cognitive Assessment | Immediately after ICU discharge and 0, 3, and 6 months after discharge
  The Montreal Cognitive Assessment (MoCA) is a brief, standardized screening tool designed to detect mild cognitive impairment. It evaluates multiple cognitive domains, including attention, executive function, memory, language, visuospatial ability, abstract thinking, calculation, and orientation. The test is scored out of 30 points, with a score of 26 or above generally considered normal.
Confusion assessment methods | Immediately after ICU discharge and 0, 3, and 6 months after discharge
  The Confusion Assessment Method (CAM) is a widely used, validated tool for the detection of delirium in clinical settings. It allows non-psychiatric clinicians to identify delirium quickly and accurately based on four key diagnostic features: (1) Acute onset and fluctuating course; (2) Inattention; (3) Disorganized thinking; (4) Altered level of consciousness. A diagnosis of delirium using CAM requires the presence of features 1 and 2, plus either feature 3 or 4.
Body weight | Immediately after ICU discharge and 0, 1, 2, 3, 4, 5, and 6 months after discharge
  Body weight refers to the total mass of an individual and is typically measured in kilograms (kg) using a calibrated digital or mechanical scale. It is a key parameter in clinical assessments, nutritional evaluations, and outcome monitoring.
Calf circumference | Immediately after ICU discharge and 0, 1, 2, 3, 4, 5, and 6 months after discharge
  Calf circumference is a simple and non-invasive anthropometric measurement used to assess muscle mass and nutritional status, particularly in older adults. Calf circumference was measured at the widest point of the non-dominant leg using a flexible, non-elastic tape measure, with participants in a seated position and knees at 90 degrees. Measurements were recorded to the nearest 0.1 cm. Cut-off values of <34 cm for men and <33 cm for women were used to identify low muscle mass, according to the AWGS 2019 criteria.
Maslach Burnout Inventory - Human Services Survey (MBI-HSS) | 0, 6, 12, 18, and 24 months after I-CARE program start
  The MBI-HSS is a widely used psychological assessment tool designed to measure burnout specifically in professionals working in human services and healthcare, such as nurses, doctors, social workers, and therapists. The survey consists of 22 items (questions). It measures three key dimensions of burnout: (1)Emotional Exhaustion; (2)Depersonalization; (3)Personal Accomplishment. Respondents rate the frequency of experiencing each feeling or attitude on a 7-point Likert scale ranging from 0 (never) to 6 (every day). Higher scores in Emotional Exhaustion and Depersonalization, along with lower scores in Personal Accomplishment, indicate greater levels of burnout.
Intention to leave | 0, 6, 12, 18, and 24 months after I-CARE program start
  Intention to leave is measured by the level of agreement with the following three statements: (1) I plan to leave my job within the next year; (2) I am actively looking for other job opportunities; (3) I want to continue working in this job. Nurses rate these statements using a 5-point Likert scale (1 = strongly disagree, 5 = strongly agree). Higher scores on the first and second statements, as well as lower scores on the third statement, indicate a higher intention to leave.
Mortality rate | 1, 2, 3, 4, 5, and 6 months after discharge
  Mortality rate is a statistical measure that represents the number of deaths in a specific population during a given period of time.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
We do not plan to share the individual participant data because sharing such data requires explicit permission from our study participants to ensure their privacy and confidentiality. Additionally, there are ethical and legal considerations regarding data protection that must be strictly followed. At this time, we prioritize safeguarding participant information and complying with applicable regulations.